CLINICAL TRIAL: NCT02236013
Title: A Phase 1 Study of ASP2215 in Combination With Induction and Consolidation Chemotherapy in Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: A Study of ASP2215 in Combination With Induction and Consolidation Chemotherapy in Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-0103
Expanded Access: NCT03070093 (Approved for marketing)
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: ASP2215; Daunorubicin; Gilteritinib; Acute Myeloid Leukemia; Idarubicin; Cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib; Idarubicin; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- ASP2215 Dose Escalation (Part 1) (Experimental): Successive dose escalation cohorts will determine the maximum tolerated dose (MTD)
  Interventions: Drug: Gilteritinib; Drug: Idarubicin; Drug: Cytarabine
- ASP2215 Dose Expansion (Part 2) (Experimental): Once the MTD has been established in Part 1, up to 20 subjects will be enrolled into an expansion cohort
  Interventions: Drug: Gilteritinib; Drug: Idarubicin; Drug: Cytarabine
- Alternative Anthracycline and Schedule (Part 3) (Experimental): In Part 3, two cohorts will be enrolled to evaluate an alternative anthracycline and ASP2215 schedule
  Interventions: Drug: Gilteritinib; Drug: Idarubicin; Drug: Cytarabine; Drug: Daunorubicin
- Continuous ASP2215 Exposure during Consolidation (Part 4) (Experimental): During Consolidation, ASP2215 will be given daily on day 1 up to day 56.
  Interventions: Drug: Gilteritinib; Drug: Idarubicin; Drug: Cytarabine; Drug: Daunorubicin

INTERVENTIONS:
Drug: Gilteritinib — Oral
  Other Names: ASP2215
Drug: Idarubicin — lyophilized powder administered intravenously
Drug: Cytarabine — solution administered intravenously
Drug: Daunorubicin — solution administered intravenously
  Arms: Alternative Anthracycline and Schedule (Part 3); Continuous ASP2215 Exposure during Consolidation (Part 4)

SUMMARY:
The purpose of this study is to describe the dose limiting toxicities (DLT) and define the maximum tolerated dose (MTD) of ASP2215 when combined with cytarabine/idarubicin or daunorubicin remission induction in a 7+3 schedule. Safety and tolerability of ASP2215 will also be evaluated. This study will also characterize the pharmacokinetics (PK) of ASP2215 when given in combination with cytarabine/idarubicin or cytarabine/daunorubicin remission induction and high-dose cytarabine (HiDAC) consolidation therapy in newly diagnosed acute myeloid leukemia as well as evaluate the effect of ASP2215 on the PK of cytarabine.

DETAILED DESCRIPTION:
This is a four-part trial. In Part 1, subjects will be enrolled to successive cohorts to determine the maximum tolerated dose (MTD). Dose escalation decision will be made based on DLTs that occur after the first dose of ASP2215 during remission induction. The treatment will consist of three distinct periods: remission induction, consolidation and maintenance.

In Part 2, subjects will be enrolled into an expansion cohort. Subjects will receive ASP2215 at the MTD established in Part 1 or recommended expansion dose, and will also receive remission induction, consolidation and maintenance therapy. The DLT observation period during the expansion cohort will be from the start of dosing of ASP2215 during the first remission induction treatment until Day 21 of the first consolidation cycle or before the start of the second consolidation cycle, whichever is sooner; as well as from the start of maintenance treatment until Day 28 of the second maintenance cycle. If testing at a dose level must be stopped, then a lower dose may be tested for remaining subjects to be enrolled.

In Part 3, two cohorts will be enrolled to evaluate an alternative anthracycline and ASP2215 schedule. During remission induction, ASP2215 dosing will begin at day 8 and continue for 14 days to day 21. Subjects will be hospitalized during remission induction therapy while receiving chemotherapy.

In cohort 3A, some subjects will be enrolled to receive 7+3 regimen consisting of cytarabine and an alternative antracycline, daunorubicin. During remission induction subjects will receive a 7+3 induction regimen consisting of daunorubicin IV infusion on days 1 through 3 and cytarabine as a continuous infusion on days 1 through 7.

In cohort 3B, some subjects will be enrolled to receive 7+3 regimen consisting of cytarabine and idarubicin at an alternative dosing schedule for ASP2215 during remission induction. During remission induction subjects will receive a 7+3 induction regimen consisting of idarubicin by IV infusion on days 1 through 3 and cytarabine as a continuous infusion on days 1 through 7.

For Part 3, if day 21 bone marrow evaluation shows residual blasts and the bone marrow is not aplastic, a second induction cycle with the same regimen will be given starting at least 7 days after last dose of ASP2215 and no later than day 35 of the first induction cycle. Consolidation and Maintenance therapy follow the same schedule and dosage outlined in Part 1.The DLT observation period for dose escalation decisions will be from the start of ASP2215 administration during the first remission induction treatment until day 42 of the last remission induction treatment cycle or before the start of the first consolidation cycle, whichever is sooner.

A subject that receives less than 80% of the intended dose of any of the study drugs during the remission induction period may be replaced.

Part 3 may be expanded for additional subjects to ensure at least some subjects are FLT3 + in each of the Alternative Anthracycline and Schedule Cohorts.

In Part 4, the effect of continuous ASP2215 exposure during consolidation will be evaluated.

During remission induction, subjects will receive a 7+3 induction regimen consisting of daunorubicin on days 1 through 3 and cytarabine as a continuous infusion on days 1 through 7. ASP2215 will be given at the designated dose, once daily starting on day 8, and continued for 14 days until day 21. If day 21 bone marrow evaluation shows residual blasts and the bone marrow is not aplastic, a second induction cycle with the same regimen will be given starting at least 7 days after last dose of ASP2215 and no later than day 35 of the first induction cycle.

Consolidation therapy will follow the same schedule and dosage outlined in Part 1 except for the ASP2215 schedule. ASP2215 will be given at the designated dose, once daily starting on day 1 up to day 56, which is the maximum number of days between each consolidation cycle.

Subjects may participate in up to 3 consolidation cycles. Maintenance therapy and posttreatment will also follow the same schedule and dosage outlined in Part 1.

The DLT observation period will be during the first consolidation cycle only. This will be from the start of ASP2215 administration (consolidation cycle 1 day 1) until consolidation cycle 1 day 56 or the next chemotherapy cycle, whichever is sooner.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of previously-untreated de novo acute myeloid leukemia (AML) according to WHO classification (2008) documented within 28 days prior to enrollment.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Subject must meet the following criteria as indicated on the clinical laboratory tests.

  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x institutional upper limit normal (ULN)
  * Total serum bilirubin ≤ 1.5 x institutional ULN
  * Serum creatinine ≤ 1.5 x institutional ULN or an estimated glomerular filtration rate (eGFR) of > 50 ml/min as calculated by the Modification of Diet in Renal Disease (MDRD) equation.
* Subject is suitable for oral administration of study drug.
* Female subject must be either:

  * Of non-child bearing potential:
  * post-menopausal (defined as at least 1 year without any menses) prior to Screening, or
  * documented surgically sterile or status post hysterectomy (at least 1 month prior to Screening)
  * Or, if of childbearing potential,
  * must agree not to try to become pregnant during the study and for 180 days after the final study drug administration, and
  * must have a negative urine pregnancy test at Screening, and
  * must use two forms of birth control* (at least one of which must be a barrier method) starting at Screening and throughout the study period and for 180 days after the final study drug administration. *Acceptable forms of birth control include:

    1. Established use of oral, injected or implanted hormonal methods of contraception.
    2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
    3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
* Female subject must not be breastfeeding at Screening or during the study period, and for 60 days after the final study drug administration.
* Female subject must not donate ova starting at Screening and throughout the study period, and for 180 days after the final study drug administration.
* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of two forms of birth control* (one of which must be a barrier method) starting at Screening and continue throughout the study period and for 120 days after the final study drug administration.
* Male subject must not donate sperm starting at Screening and throughout the study period and for 120 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while on treatment.

Exclusion Criteria:

* Subject was diagnosed as acute promyelocytic leukemia (APL) or AML with good risk cytogenetics; t(8;21), inv(16) or t(16;16). (Subjects with pending cytogenetics that require treatment may enroll. Any subject that is found to have good risk cytogenetics after initiation of treatment will discontinue ASP2215 and be taken off trial).
* Subject has BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
* Subject has active malignant tumors other than AML or myelodysplastic syndrome (MDS).
* Subject has received previous therapy for AML, with the exception of the following:

  * Emergency leukapheresis;
  * Emergency treatment for hyperleukocytosis with hydroxyurea for ≤ 10 days;
  * Preemptive treatment with retinoic acid prior to exclusion of APL ≤ 7 days;
  * Growth factor or cytokine support;
  * Steroids for the treatment of hypersensitivity or transfusion reactions.
* Subject has clinically active central nervous system leukemia.
* Subject has disseminated intravascular coagulation abnormality (DIC).
* Subject has had major surgery within 4 weeks prior to the first study dose.
* Subject has radiation therapy within 4 weeks prior to the first study dose.
* Subject has congestive heart failure New York Heart Association (NYHA) class 3 or 4, or subject with a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram performed within 3 months prior to study entry results in a left ventricular ejection fraction that is ≥ 45%.
* Subject requires treatment with concomitant drugs that are strong inducers of cytochrome P450 (CYP)3A.
* Subject requires treatment with concomitant drugs that are strong inhibitors or inducers of P glycoprotein (P-gp) with the exception of drugs that are considered absolutely essential for the care of the subject.
* Subject requires treatment with concomitant drugs that target serotonin 5HT1R or 5HT2BR receptors or sigma nonspecific receptor with the exception of drugs that are considered absolutely essential for the care of the subject.
* Subject has an active uncontrolled infection.
* Subject is known to have human immunodeficiency virus infection.
* Subject has active hepatitis B or C, or other active hepatic disorder.
* Subject has any condition which makes the subject unsuitable for study participation (e.g. ophthalmic conditions such as advanced cataracts).
* Subject has Fridericia-corrected QT interval (QTcF) > 450 ms at Screening based on central reading.
* Subject has Long corrected QT interval (QTc) Syndrome at Screening.
* Subject has hypokalemia and hypomagnesemia at Screening (defined as values below institutional lower limit of normal [LLN]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01-07 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by development of dose limiting toxicities, adverse events, and define maximum tolerated dose (MTD) | up to 2.5 years after start of the treatment

SECONDARY OUTCOMES:
Pharmacokinetics profile of ASP2215: AUC24, Cmax, Ctrough and tmax | Days 8, 11, 17, and 28 for remission induction and Days 1, 2, and 15 for consolidation
  Area under the curve at 24 hours (AUC24), maximum concentration (Cmax), minimum concentration (Ctrough), and time after dosing when Cmax occurs (tmax)
Pharmacokinetics of cytarabine: Css | Days 3 and 8
  Steady state concentration (Css)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (10):
- United States (10):
  - Site US10003, Los Angeles, California
  - Site US10013, New Haven, Connecticut
  - Site US10004, Chicago, Illinois
  - Site US10009, Westwood, Kansas
  - Site US10001, Baltimore, Maryland
  - Site US10002, New York, New York
  - Site US10014, Cleveland, Ohio
  - Site US10019, Oklahoma City, Oklahoma
  - Site US10006, Philadelphia, Pennsylvania
  - Site US10010, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Pratz KW, Cherry M, Altman JK, Cooper BW, Podoltsev NA, Cruz JC, Lin TL, Schiller GJ, Jurcic JG, Asch A, Wu R, Hill JE, Gill SC, James AJ, Rich ES, Hasabou N, Perl AE, Levis MJ. Gilteritinib in Combination With Induction and Consolidation Chemotherapy and as Maintenance Therapy: A Phase IB Study in Patients With Newly Diagnosed AML. J Clin Oncol. 2023 Sep 10;41(26):4236-4246. doi: 10.1200/JCO.22.02721. Epub 2023 Jun 28. PMID 37379495